CLINICAL TRIAL: NCT01469325
Title: Effectiveness of of Sequential Left Prefrontal Repetitive Transcranial Magnetic Stimulation, With High Frequency, for Treatment-Resistant Depression, in TMS Unit, Neurcognitive Lab, Iranian National Center for Addiction Studies (INCAS), in 2011. A Randomized, Controlled Trial.
Brief Title: Sequential Left Prefrontal Repetitive Transcranial Magnetic Stimulation, With High Frequency, for Treatment-Resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Khazaeipour, Principal Investigator, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 90-03-49-14937; 90-03-49-14937
Record Dates: First submitted 2011-11-02; First posted 2011-11-10 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Treatment-Resistant Depression Disease
Keywords: Repetitive Transcranial Magnetic Stimulation; Depression; left prefrontal
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Repetitive Transcranial Magnetic Stimulation (Active Comparator): We deliver rTMS to the left prefrontal cortex at 120% motor threshold (10 Hz, 4-second train duration, and 26-second intertrain interval) for 37.5 minutes (3000 pulses per session) using a figure-eight solid-core coil.
  Interventions: Other: Repetitive Transcranial Magnetic Stimulation
- Sham rTMS (Sham Comparator): Sham rTMS using a similar coil with a metal insert blocking the magnetic field and scalp electrodes that delivered matched somatosensory sensations.
  Interventions: Other: Sham rTMS

INTERVENTIONS:
Other: Repetitive Transcranial Magnetic Stimulation — We deliver rTMS to the left prefrontal cortex at 120% motor threshold (10 Hz, 4-second train duration, and 26-second intertrain interval) for 37.5 minutes (3000 pulses per session) using a figure-eight solid-core coil
  Arms: Repetitive Transcranial Magnetic Stimulation
Other: Sham rTMS — Sham rTMS using a similar coil with a metal insert blocking the magnetic field and scalp electrodes that delivered matched somatosensory sensations.
  Arms: Sham rTMS

SUMMARY:
Sequential left prefrontal Repetitive Transcranial Magnetic Stimulation (rTMS), with high frequency, for Treatment-Resistant Depression have been shown to have antidepressant effects. but doubts remain about the magnitude of previously demonstrated treatment effects.The aim of this study is To test whether daily weekday left prefrontal rTMS safely and effectively treats Resistant Depression disorder compared to sham controls.

DETAILED DESCRIPTION:
Design:

Prospective, randomized, active sham-controlled (1:1 randomization), duration-adaptive design with 3 weeks of daily weekday treatment (fixed-dose phase) followed by continued blinded treatment for up to another 3 weeks in improvers.

Setting:

University psychiatric hospitals in Tehran including Roozbeh Hospital, Rasool Hospital and Imam Hossein General Hospital will refer clients to Iranian National Center for Addiction Studies, Tehran University of Medical Sciences.

Patients:

About 60 patients with unipolar nonpsychotic major depressive disorder, according to DSM-IV, resistant to treatment.

INTERVENTION:

We delivered rTMS to the left prefrontal cortex at 120% motor threshold (10 Hz, 4-second train duration, and 26-second intertrain interval) for 37.5 minutes (3000 pulses per session) using a figure-eight solid-core coil. Sham rTMS used a similar coil with a metal insert blocking the magnetic field and scalp electrodes that delivered matched somatosensory sensations.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of major depression
* Resistance to treatment as defined by the insufficient clinical benefit to at least one adequate medication trials

Exclusion Criteria:

* Other current Axis I disorders (except simple phobia and nicotine addiction)
* Personal or close family history of seizure disorder
* Ferromagnetic material in body or close to head
* Neurologic disorder
* Pregnancy
* Taking medications known to lower seizure threshold (eg, theophylline)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
change (decrease) of depression according to Hamilton, Beck, BPRS questionnaires. | 3 week
  The primary outcome measure for the study was score on the MADRS. The patients were assessed with the MADRS, the 17-item version of the Hamilton Depression Rating Scale (HAM-D), the Beck Depression Inventory (BDI), the Brief Psychiatric Rating Scale (BPRS), the CORE Rating of Psychomotor Disturbance (16), and the Global Assessment of Functioning (GAF) Scale (DSM-IVTR).

CONTACTS AND LOCATIONS:
Locations (1):
- Iranian National Center for Addiction Studies, Tehran, Tehran Province, Iran